CLINICAL TRIAL: NCT03651999
Title: Influence of the "Atelier du rêve" (Dream Workshop) on the Quality of Falling Asleep in the Operating Room.
Acronym: REVA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: REVA
Record Dates: First submitted 2018-08-01; First posted 2018-08-29 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dream workshop: After consultation with the pediatric surgeon or the anesthesiologist, parents and children are invited to meet the nurse anesthetist, in a room dedicated to this purpose and specially designed to accommodate children; they will find a playmobil model, photographs of the patient circuit as well as different games or activities that can be performed during induction; The nurse anesthetist explains the hospitalization process and will help them to choose a pleasant dream, a perfume adapted to their taste, a distraction adapted to their age (animated book, soap bubbles, favorite song ...); the child will be able to customize his mask and choose the blanket he wants to take along; the most recalcitrant or special sites (autism, long-term hospitalization) will be able to be accompanied by a parent during sleep
  Interventions: Other: participation in a workshop: "dream workshop" animated by a nurse anesthesist
- control: No "dream workshop"

INTERVENTIONS:
Other: participation in a workshop: "dream workshop" animated by a nurse anesthesist — After consultation with the pediatric surgeon or the anesthesiologist, parents and children are invited to meet the nurse, in a room dedicated to this purpose and specially designed to accommodate children; they will find a playmobil model, photographs of the patient circuit as well as different games or activities that can be performed during induction; the nurse anesthetist will take care to explain to them the progress of the hospitalization and help them to choose a pleasant dream, a perfume adapted to their taste, a distraction adapted to their age (animated book, soap bubbles, favorite song ...) ; he can customize his mask and choose the blanket he wants to take; the most recalcitrant or special sites (autism, long-term hospitalization) will be able to be accompanied by a parent during sleep
  Groups: dream workshop

SUMMARY:
A "dream workshop" is organized for the children by nurses specialized in anesthesia in the CHI Creteil. During this workshop, the anesthesia process is explained to the children using games, drawings, songs, etc. The impact of this workshop on the child stress and acceptance of the mask during induction is studied in this research.

DETAILED DESCRIPTION:
For more than two years, nurse anesthetists have developed a personalized treatment of children who will be asleep using the theoretical bases of hypnosis in children and distraction, in order to improve the conditions of falling asleep, especially by promoting the acceptance of the mask during inhalation induction, or by preparing it for an Intra Venous induction, if it so desires or if it is obligatory.

Indeed, the announcement of a surgical intervention is sometimes experienced as a real emotional shock by the parents and / or the child, whatever the gravity or the stake of the surgical gesture. To all this is added the phobic fear of anesthesia and all conditions are met to generate a climate of maximum stress. The work of nurse anesthesists prior to this surgical procedure was to establish a relationship of trust with the child through this "dream workshop", to restore a more serene climate.

Thus, is it the idea of this "workshop of the dream", allowing thanks to the imagination of the child, to recreate a universe of confidence full of colors, songs and perfume ...

After consultation with the pediatric surgeon or the anesthesiologist, parents and children are invited to meet nurse anesthesists, if they wish, in a room dedicated to this purpose and specially designed to accommodate children; they will find a playmobil model, photographs of the patient circuit as well as different games or activities that can be performed during induction; the nurse anesthetist will take care to explain to them the progress of the hospitalization and help them to choose a pleasant dream, a perfume adapted to their taste, a distraction adapted to their age (animated book, soap bubbles, favorite song ...) ; he can customize his mask and choose the blanket he wants to take; the most recalcitrant or special sites (autism, long-term hospitalization) will be able to be accompanied by a parent during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Children who need an ambulatory surgery
* benefiting from a health care insurance

Exclusion Criteria:

* surgery planned in another hospital
* hospitalized children
* refusal to participate

Ages: 3 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: children from 3 to 8 years old planned ambulatory surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Acceptance or not acceptance of the mask in the operating room | day of planned surgery
  evaluated by the operating nurse

SECONDARY OUTCOMES:
Paediatric Anaesthesia Emergence Delirium score | day of planned surgery
Yale Preoperative Anxiety Scale | day of planned surgery
Visual analogic anxiety score | day of planned surgery
  on a 0 to 10 scale
Face Legs Activity Cry Consolability | 1h post planned surgery
  post-surgery pain in the recovery room
Post Hospitalization Behavior Questionnaire | day 1 post planned surgery
Post Hospitalization Behavior Questionnaire | day 7 post planned surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lebourdiec, Principal Investigator — CHI CRETEIL
Locations (1):
- CHi Creteil, Créteil, France